CLINICAL TRIAL: NCT04762615
Title: Impact of the Immunosuppressive Treatment, X-ray Exposition and Renal Pathology on Ovarian Reserve in Young Women
Brief Title: Impact of Underlying Renal Disease and Immunosuppressive Regimen on Ovarian Reserve in Renal Patients
Status: Completed | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 451/2018
Record Dates: First submitted 2021-02-02; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-12

CONDITIONS: Anti-Mullerian Hormone Deficiency; Immunosuppression; Ovarian Reserve; X-rays; Effects
Keywords: AMH; Immunosuppression; Ovarian Reserve; X-Ray effects

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with renal pathology treated with immunosuppressive drugs: Female in reproductive age suffering from renal disease that is or was previously treated with immunosuppressive drugs
  Interventions: Diagnostic Test: AMH level measurement
- Patients with renal pathology without treatment: Control group
  Interventions: Diagnostic Test: AMH level measurement
- Patients after renal transplantation taking immunosuppressive drugs: Female in reproductive age after renal transplantation taking immunosuppressive drugs
  Interventions: Diagnostic Test: AMH level measurement

INTERVENTIONS:
Diagnostic Test: AMH level measurement — AMH level measurement using ELISA test from blood samples

SUMMARY:
Aging, renal pathology (eg SLE, ADPKD), X-ray exposition and pharmacological treatments, especially previous strong immunosuppression, may negatively influence the ovarian reserve in childbearing age women. Anti-Müllerian hormone (AMH) is regarded as biomarker for ovarian reserve.

Every female with renal disease regularly menstruating that met exclusion criteria could have participated. The aim was to assess ovarian reserve in female patients with normal menstrual cycle and kidney disease, including kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Conscious written approval
* Autoimmunological disorder with kidneys affection/ kidney transplant recipient- Regular menstrual cycles
* Age above 18 years old

Exclusion Criteria:

* Irregular menstrual cycles
* Menopause
* PCOS
* Chemiotherapy or radiotherapy in the past
* Surgical interventions within ovaries
* Hypogonadotropic hypogonadism
* Folliculoma
* Age under 18 years old

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female patients
Study Population: Regularly menstruating female patients suffering from renal pathology or after renal transplantation
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
To compare AMH levels between three groups | 1 day
  Serum AMH levels [ng/ml] measured using ELISA and compared between three groups
Potential impact of X-ray exposition on ovarian reserve | 1 day
  Analysis of the impact of X-ray exposition [mSv] on AMH serum level [ng/ml]
Potential impact of antiproliferative drugs on ovarian reserve | 1 day
  Analysis of the impact of antiproliferative drugs on AMH serum level [ng/ml]
Potential impact of underlying kidney disease on ovarian reserve | 1 day
  Analysis of the impact of underlying kidney disease (including SLE) on AMH serum level [ng/ml]

CONTACTS AND LOCATIONS:
Overall Officials: Julia Rasała, MD, Principal Investigator — Wroclaw Medical University
Locations (1):
- Nephrology and Transplantation Clinic University Hospital in Wrocław, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No